CLINICAL TRIAL: NCT00004843
Title: A Randomized Study of Surgery vs No Surgery in Patients With Mild Asymptomatic
Brief Title: A Randomized Study of Surgery vs No Surgery in Patients With Mild Asymptomatic Primary Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Henry Ford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 199/13926; R01DK043858 (NIH)
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hyperparathyroidism
Keywords: disease-related problem/condition; endocrine disorders; hyperparathyroidism; quality of life; rare disease
MeSH Terms: conditions — Hyperparathyroidism; Endocrine System Diseases; Rare Diseases | interventions — Parathyroidectomy; Observation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parathyroidectomy (Experimental)
  Interventions: Procedure: parathyroidectomy
- Observation (Active Comparator)
  Interventions: Other: Observation

INTERVENTIONS:
Procedure: parathyroidectomy — Standard parathyroidectomy with a bilateral approach
  Arms: Parathyroidectomy
Other: Observation — Usual care
  Arms: Observation

SUMMARY:
OBJECTIVES: I. Assess the efficacy of surgery vs no surgery in patients with mild asymptomatic primary hyperparathyroidism.

II. Assess the quality of life, morbidity, and mortality of these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are stratified by gender. Patients are randomized to receive surgery or follow up without surgery.

Patients receive parathyroidectomy (current standard care) or long term follow up without parathyroidectomy.

Quality of life is assessed before the study and then every 6 months. All patients are followed every 6 months until death.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically diagnosed mild asymptomatic primary hyperparathyroidism Persistent albumin adjusted serum calcium between 10.1-11.5 mg/dL for at least 3 months Intact parathyroid hormone greater than 20 pg/mL No other cause for hypercalcemia No family history of primary hyperparathyroidism, primary endocrine neoplasia, or hypocalciuric hypercalcemia Bone mineral density of the forearm no greater than 2.0 SD units below the expected value for sex, age, and race No phalangeal subperiosteal resorption on hand x-rays --Prior/Concurrent Therapy-- Radiotherapy: No history of childhood irradiation to head and neck Surgery: No thyroid disease requiring surgical intervention Other: No prior glucocorticoid or anticonvulsant drug therapy Concurrent thiazide diuretic therapy for hypertension must be changed to nonthiazides --Patient Characteristics-- Menopausal status: At least 5 years postmenopausal Renal: At least 2 years since prior nephrolithiasis Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 70% (age adjusted) Cardiovascular: No unexpected finding on echocardiogram that will interfere with surgical intervention Other: Living within 150 mile radius of downtown Detroit No concurrent participation in other clinical trials No concurrent polyuria, polydipsia, anorexia, nausea, or vomiting At least 12 months since prior pancreatitis No concurrent symptomatic peptic ulcer disease No objective muscle weakness No history of nontraumatic vertebral or hip fractures No vertebral compression fractures No urolithiasis on x-ray of abdomen

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1997-04 (Actual); Primary Completion 1999-03-30 (Actual); Study Completion 1999-03-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 2 years
  Change in 9 SF 36 scores

CONTACTS AND LOCATIONS:
Overall Officials: D. Sudhaker Rao, Study Chair — Henry Ford Hospital

REFERENCES:
- [Result] Talpos GB, Bone HG 3rd, Kleerekoper M, Phillips ER, Alam M, Honasoge M, Divine GW, Rao DS. Randomized trial of parathyroidectomy in mild asymptomatic primary hyperparathyroidism: patient description and effects on the SF-36 health survey. Surgery. 2000 Dec;128(6):1013-20;discussion 1020-1. doi: 10.1067/msy.2000.110844. PMID 11114637